CLINICAL TRIAL: NCT02159703
Title: A Single-arm Phase II Study of Post-Transoral Robotic Surgery (TORS) Alone to the Primary Tumor Site and Selective Neck Dissection (SND) Followed by Adjuvant Radiation Therapy (+/- Chemotherapy) to the Regional Nodes for Advanced Stage, Human Papilloma Virus (HPV) Positive, Oropharyngeal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Diagnostic
Other Study IDs: UPCC 40313
Record Dates: First submitted 2014-06-06; First posted 2014-06-10 (Estimated); Results first posted 2019-11-21 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Oropharyngeal Cancer
Keywords: T1-2 N2 M0,; stage IVa SCCA; oropharynx; negative for PNI,; negative surgical margins
MeSH Terms: conditions — Oropharyngeal Neoplasms; Margins of Excision

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm Phase 2 (Experimental)
  Interventions: Procedure: TORS; Radiation: Adjuvant Radiation Therapy

INTERVENTIONS:
Procedure: TORS
Radiation: Adjuvant Radiation Therapy

SUMMARY:
To determine 2-year local (primary tumor site) control and toxicity rates in patients receiving adjuvant RT post-TORS, omitting the primary tumor bed, in patients with completely resected, HPV-positive SCCA of the oropharynx.

To determine acute and long-term toxicity rates in patients receiving adjuvant RT post-TORS, omitting the primary tumor bed, in patients with completely resected, HPV-positive SCCA of the oropharynx.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older Histologically confirmed diagnosis of squamous cell carcinoma of the oropharynx, stage IVa, p16-positive on immunohistochemistry Pathologic T1 or T2 disease, resected with negative margins ( 2mm) Pathologic N2a, N2b, or N2c disease ECOG Performance Status 0-1
* Patients must sign an informed consent document that indicates they are aware of the investigational nature of the treatment in this protocol as well as the potential risks and benefits - - - Ability to understand and the willingness to provide written informed consent

Exclusion Criteria

* Prior radiation therapy to the head and neck Prior chemotherapy within the past 5 years Presence of T3 or T4 disease Presence of close (2 mm) or positive margins PNI on TORS resection of the primary cancer Presence of N0 or N1 disease in neck dissection Presence of distant metastatic (M1) disease
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, connective tissue disease or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-02; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Lin, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Swisher-McClure S, Lukens JN, Aggarwal C, Ahn P, Basu D, Bauml JM, Brody R, Chalian A, Cohen RB, Fotouhi-Ghiam A, Geiger G, Gershowitz J, Livolsi V, Mitra N, Montone K, Newman J, Ojerholm E, O'Malley B Jr, Rajasekaran K, Tan E, Weinstein G, Lin A. A Phase 2 Trial of Alternative Volumes of Oropharyngeal Irradiation for De-intensification (AVOID): Omission of the Resected Primary Tumor Bed After Transoral Robotic Surgery for Human Papilloma Virus-Related Squamous Cell Carcinoma of the Oropharynx. Int J Radiat Oncol Biol Phys. 2020 Mar 15;106(4):725-732. doi: 10.1016/j.ijrobp.2019.11.021. Epub 2019 Nov 27. PMID 31785337

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm Phase 2: Post-Transoral Robotic Surgery (TORS) Alone to the Primary Tumor Site and Selective Neck Dissection (SND) Followed by Adjuvant Radiation Therapy (+/- Chemotherapy)
Period: Overall Study
Arm/Group | Single Arm Phase 2
Started | 60
Completed | 60
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Single Arm Phase 2: TORS
  Adjuvant Radiation Therapy
Arm/Group | Single Arm Phase 2
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 45
  >=65 years | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.51 (9.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 60
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 58
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Local Control
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Single Arm Phase 2
Number analyzed (Participants) | 60
percentage of patients | 97.9 [86.1 to 99.7]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Single Arm Phase 2
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 18/60
Other Adverse Events (participants affected / at risk) | 43/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm Phase 2 (N=60)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dermatitis radiation (Injury, poisoning and procedural complications) | 8 (8)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Esophageal pain (Gastrointestinal disorders) | 1 (1)
Other Gastrointestinal disorders (Gastrointestinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm Phase 2 (N=60)
Alopecia (Skin and subcutaneous tissue disorders) | 18 (18)
Anorexia (Metabolism and nutrition disorders) | 19 (28)
Anxiety (Psychiatric disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Constipation (Gastrointestinal disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Depression (Psychiatric disorders) | 2 (2)
Dermatitits radiation (Injury, poisoning and procedural complications) | 39 (79)
Dizziness (Nervous system disorders) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 33 (44)
Dysgeusia (Nervous system disorders) | 40 (73)
Dysphagia (Gastrointestinal disorders) | 23 (36)
Other Ear and labyrinth disorders (Ear and labyrinth disorders) | 1 (1)
Edema face (General disorders) | 2 (2)
Esophageal pain (Gastrointestinal disorders) | 12 (17)
Fatigue (General disorders) | 26 (34)
Other Gastrointestinal disorders (Gastrointestinal disorders) | 3 (3)
Other General disorders and administration site conditions (General disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hypothyroidism (Endocrine disorders) | 4 (4)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Lip pain (Gastrointestinal disorders) | 1 (1)
Lymphedema (Vascular disorders) | 20 (24)
Mucosal infection (Infections and infestations) | 11 (25)
Mucositis oral (Gastrointestinal disorders) | 18 (24)
Other Musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3)
Neck edema (General disorders) | 4 (4)
Other Nervous system disorders (Nervous system disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 2 (2)
Pain (General disorders) | 2 (2)
Salivary duct inflammation (Gastrointestinal disorders) | 28 (38)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Superficial soft tissue fibrosis (Musculoskeletal and connective tissue disorders) | 11 (11)
Trismus (Musculoskeletal and connective tissue disorders) | 2 (2)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 18 (22)
Vomiting (Gastrointestinal disorders) | 1 (1)
Weight loss (Investigations) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-24): https://cdn.clinicaltrials.gov/large-docs/03/NCT02159703/Prot_SAP_000.pdf